CLINICAL TRIAL: NCT01258842
Title: Double-blind, Randomized, Placebo-controlled Trial of the Effects of Prophylactic Bifidobacterium Lactis HN019 Supplementation on the Incidence of Influenza Infection in Healthy Adults
Brief Title: Bifidobacterium Lactis HN019 Supplementation for Prevention of Influenza Infection in Healthy Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fonterra Research Centre (Industry)
Collaborators: Danisco (Industry); Sprim Advanced Life Sciences (Other)
Responsible Party: Pramod Gopral, PhD, Fonterra Research Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 10-SBUS-6-FON-02
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Influenza
Keywords: Influenza; Prevention; Probiotic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B. lactis HN019 (Experimental)
  Interventions: Dietary Supplement: Bifidobacterium lactis HN019
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium lactis HN019 — B. lactis HN019 (5 billion cfu / day) sachet, consumed once per day for 12 weeks
  Arms: B. lactis HN019
Dietary Supplement: Placebo — Placebo sachet, consumed once per day for 12 weeks
  Arms: Placebo

SUMMARY:
To determine if prophylactic supplementation with B. lactis HN019 reduces the risk of developing physician- and laboratory-confirmed influenza infection at any time during the 12-week supplementation period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy free-living men and women aged 18 to 60 years
* Body mass index between 18.5 and 29.9 kg/m2 (encompasses normal weight and overweight)
* Subject owns a refrigerator and is willing to keep study product refrigerated at all times
* Ability of the participant (in the investigator's opinion) to comprehend the full nature and purpose of the study, including possible risks and side effects
* Consent to the study and willing to comply with study product and methods

Exclusion Criteria:

* Influenza vaccination in last 6 months, or any other vaccination in previous 15 days
* Clinically significant underlying systemic illness that may preclude the subject's ability to complete the trial
* Chronic nasal, laryngeal, pleural, or respiratory condition that could mimic or obscure symptoms of influenza (e.g. chronic allergic rhinitis, asthma, COPD, as determined by medical history and baseline physical examination)
* Chronic use of medication(s) that could suppress or prevent flu-like symptoms (eg, antihistamines, cough medicines; echinacea, high-dose vitamin C)
* Use of medication(s) within the previous 3 months that affect immune response (eg, antibiotics)
* Contraindication to dairy products or any other substance in the study product (eg, lactose intolerance)
* History of alcohol, drug, or medication abuse
* Pregnant or lactating female, or pregnancy planned during study period
* Daily consumption of probiotics, prebiotics, fermented milk, and/or yogurt within 3 months of screening
* Participation in another study with any investigational product within 3 months of screening
* Investigator believes that the participant may be uncooperative and/or noncompliant, and should therefore not participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 426 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Influenza infection | 12 weeks
  Incidence of physician- and laboratory-confirmed influenza infection at any time during the 12-week supplementation period

SECONDARY OUTCOMES:
Symptom duration | 12 weeks
Symptom severity | 12 weeks
Adverse event incidence | 12 weeks
  The proportion of subjects that reports at least one adverse event (regardless of cause) during the study

CONTACTS AND LOCATIONS:
Overall Officials: Mario Clerici, MD, Principal Investigator — Milano University Medical School; Emilio Clementi, Principal Investigator — University of Milan
Locations (2):
- United States (2):
  - Clinical Research of South Florida, Coral Gables, Florida
  - Remedica, LLC, Rochester, Michigan